CLINICAL TRIAL: NCT03496155
Title: A Pilot Efficacy and Implementation Study of the Strengths Intervention Project
Acronym: SIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: John Templeton Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 18-014922
Record Dates: First submitted 2018-03-21; First posted 2018-04-12 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Parent-Child Relations; Parenting; Adolescent Behavior; Communication
Keywords: parent-teen communication; teen strengths; adolescence
MeSH Terms: conditions — Adolescent Behavior; Communication

STUDY DESIGN:
Intervention Model Description: Treatment groups receive intervention and control groups receive usual care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Intervention Group (Arm 1- Main) (Experimental): Will receive the "Build Your Teen's Strengths" educational pamphlet, health coaching sessions, and provider endorsement.
  Interventions: Behavioral: Build and Support Your Teen's Strengths
- Control Group (Arm 1- Main) (No Intervention): Will receive usual care at well-child visit.
- Intervention Group (Arm 1-asthma subgroup) (Experimental): Will receive the "Build Your Teen's Strengths" educational pamphlet, health coaching sessions, and provider endorsement.
  Interventions: Behavioral: Build and Support Your Teen's Strengths
- Control Group (Arm 1-asthma subgroup) (No Intervention): Will receive usual care at well-child visit.
- Control Group (Arm 2) (No Intervention): Convenience sample used for a post-hoc, exploratory analysis. Will receive usual care at well-child visit.

INTERVENTIONS:
Behavioral: Build and Support Your Teen's Strengths — This is a clinic based psychoeducational intervention for adolescent patients and their parents to improve parent-teen communication about teen strengths. The intervention is designed, if possible, to coincide with the adolescent patients' well-child visits and consists of the following components: (1) In-person or over the phone orientation session with a trained health coach and parent, (2) Distribution of psychoeducational materials to the parent, (3) Endorsement and delivery of key messages from the health care provider, and (4) "Booster" phone call placed by the health coach.
  Arms: Intervention Group (Arm 1- Main); Intervention Group (Arm 1-asthma subgroup)

SUMMARY:
The purpose of this study is to test a strengths-based intervention to be delivered in a primary care setting with adolescents and a parent. Investigators want to find out if the intervention can help parents and teens communicate. Specifically Investigators want to see if they can help parents and teens identify and build teen's strengths. Half the dyads will receive the educational materials in conjunction with their teen's well-child visit, while the other half will receive usual care at the well-child visit and receive the educational materials at the end of the study. Additionally, Investigators expect that a strengths-based intervention may also impact adherence to treatment in youth with a chronic illness. As such, Investigators will include a subgroup of teenagers diagnosed with asthma in this study, to assess whether the strengths-based intervention that the Investigators developed has an impact on adherence.

DETAILED DESCRIPTION:
Recent research suggests that parents and adolescents report an interest in doctors facilitating increased parent-teen communication about teen strengths. However, little research focuses on how to address this need in a primary care setting. Content from subject matter experts along with data gathered from parents and teens were used to develop a novel strengths-based intervention to be tested in primary care.

The study intervention being examined is called the Strengths Intervention Project and includes a written pamphlet, a guided discussion activity, in-person/phone health coaching, and in-person or mailed health care provider endorsement and key messaging. Measures will be collected at baseline pre-intervention (T1), in clinic or over the phone at the time of the intervention (T2), approximately two weeks post-intervention (T3), and approximately 2 months post-intervention (T4). Daily diaries will also be utilized twice to gather data pre- and post- intervention. We will measure feasibility of clinic implementation of intervention, as well as influence of intervention on parent-teen communication and adolescent outcomes.

ELIGIBILITY:
Adolescent Criteria:

Inclusion Criteria:

1. Teens age 13 to 15 years at the time of their upcoming well-child visit (Arm 1) OR Teens age 13 to 15 years at the time of their last well-child visit (Arm 2)
2. Children's Hospital of Philadelphia (CHOP) primary care patient (Arm 1 and 2)
3. Scheduled for a well-child visit that parent and teen both plan to attend (Arm 1) OR Attended a well-child visit with parent (Arm 2)
4. Diagnosed with Asthma > year (asthma subgroup; Arm 1 only)
5. Prescribed a controller medication year-round (asthma subgroup; Arm 1 only)
6. Adolescent has their own email account to complete electronic surveys (Arm 1 and 2)

Exclusion Criteria:

1. Not fluent in written or spoken English (Arm 1 and 2)
2. Attending a new patient well-child visit (Arm 1) OR attended a new patient well-child visit (Arm 2)
3. Presence of developmental delay or pervasive developmental disorder that requires special education services (Arm 1 and 2)
4. Psychiatric hospitalization of the adolescent in the past year (Arm 1 and 2)
5. Participated in studies: CHOP IRB # 15-011732 and/or CHOP IRB # 17-013895 (Arm 1 and 2)
6. Adolescent has sibling enrolled in (IRB 18-014922) (Arm 1 and 2)

Parent Criteria:

Inclusion Criteria:

1. Parent or legal guardian of a teen age 13 to 15 years at their upcoming well-child visit at a CHOP primary care practice (Arm 1) OR Parent or legal guardian of a teen age 13 to 15 years at their recent well-child visit at a CHOP primary care practice (Arm 2)
2. Parent has their own email account to complete electronic surveys (Arm 1 and 2)

Exclusion Criteria:

1. Not fluent in written or spoken English (Arm 1 and 2)
2. Participated in studies: CHOP IRB # 15-011732 and/or CHOP IRB # 17-013895 (Arm 1 and 2)

Ages: 13 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 174 (Actual)
Dates: Start 2018-05-04 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Change in Beliefs about Adolescents | Baseline (T1) and 2-months (T4)
  26 items (parents only); Likert scale (1= very unlikely; 7= very, very likely)
Change in Parent-Adolescent Communication (PACS) | Baseline (T1) and 2-months (T4)
  20 items (parent and teens); Likert scale (1= strongly disagree; 5= strongly agree)
Change in Confidence in exploring and using adolescent's strengths | Baseline (T1) and 2-months (T4)
  15 items (parents and teens); Likert scale (1=strongly disagree; 5= strongly agree)
Feasibility of consent rates | 9 months
  Feasibility will be demonstrated by consent rates ≥60%
Feasibility of intervention implementation | 1 month
  Completion of core intervention components ≥ 70%.
Parent and adolescent acceptability of intervention materials | 2-weeks post intervention (T3)
  Adolescent and parent acceptability ratings ≥80%. Investigators will also elicit open-ended feedback.
Parent and adolescent acceptability of intervention materials (additional) | 2-months post intervention (T4)
  2 items (parents and teens); Yes/No/Not sure and Likert scale (1=very likely; 5 very unlikely)
Provider acceptability of intervention | 9 months
  Provider acceptability ratings ≥80%. Investigators will also elicit open-ended feedback.

SECONDARY OUTCOMES:
Change in Psychological well-being using the Flourishing Scale | Baseline (T1) and 2-months (T4)
  Measure of psychological well-being. 8 items (parents and teens). (Likert scale 1= Strongly disagree; 2= Disagree; 3= Slightly disagree; 4= Mixed or neither agree nor disagree; 5= Slightly agree; 6= Agree; 7= Strongly agree). Score will be summed for range of 8 (Strong Disagreement with all items) to 56 (Strong Agreement with items). High scores signify that respondents view themselves in positive terms in important areas of functioning.
Change in Adherence to inhaled controller medication use | Baseline (T1) and 2-months (T4)
  2-items about adherence to inhaled controller medication use (parent and teen) will be assessed using the Visual analog scale (0-10).

CONTACTS AND LOCATIONS:
Overall Officials: Victoria A Miller, PhD, Principal Investigator — Children's Hospital of Phiadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ford CA, Cheek C, Culhane J, Fishman J, Mathew L, Salek EC, Webb D, Jaccard J. Parent and Adolescent Interest in Receiving Adolescent Health Communication Information From Primary Care Clinicians. J Adolesc Health. 2016 Aug;59(2):154-61. doi: 10.1016/j.jadohealth.2016.03.001. Epub 2016 Apr 14. PMID 27151760
- [Background] Jaccard J, Dodge T, Dittus P. Parent-adolescent communication about sex and birth control: a conceptual framework. New Dir Child Adolesc Dev. 2002 Fall;(97):9-41. doi: 10.1002/cd.48. No abstract available. PMID 14964942
- [Background] Elster AB, Kuznets NJ. AMA Guidelines for Adolescent Preventive Services (GAPS): Recommendations and Rationale. Baltimore: Williams & Wilkins; 1994.
- [Background] Hagan J, Shaw J, PM Duncan PM e. Bright Futures: Guidelines for Health Supervision of Infants, Children, and Adolescents 4th ed. Elk Grove Village, IL: American Academy of Pediatrics; 2017.
- [Background] Ford CA, Davenport AF, Meier A, McRee AL. Partnerships between parents and health care professionals to improve adolescent health. J Adolesc Health. 2011 Jul;49(1):53-7. doi: 10.1016/j.jadohealth.2010.10.004. Epub 2011 Mar 12. PMID 21700157
- [Background] Duncan PM, Garcia AC, Frankowski BL, Carey PA, Kallock EA, Dixon RD, Shaw JS. Inspiring healthy adolescent choices: a rationale for and guide to strength promotion in primary care. J Adolesc Health. 2007 Dec;41(6):525-35. doi: 10.1016/j.jadohealth.2007.05.024. Epub 2007 Aug 29. PMID 18023780
- [Background] Catalano RF, Berglund ML, Ryan JAM, et al. Positive youth development in the United States: research findings on evaluations of positive youth development programs. Ann Am Acad Pol Soc Sci 2004;591:98 -125.
- [Background] Mangione-Smith R, DeCristofaro AH, Setodji CM, Keesey J, Klein DJ, Adams JL, Schuster MA, McGlynn EA. The quality of ambulatory care delivered to children in the United States. N Engl J Med. 2007 Oct 11;357(15):1515-23. doi: 10.1056/NEJMsa064637. PMID 17928599
- [Background] Hammig B, Jozkowski K. Health Education Counseling During Pediatric Well-Child Visits in Physicians' Office Settings. Clin Pediatr (Phila). 2015 Jul;54(8):752-8. doi: 10.1177/0009922815584943. Epub 2015 Apr 29. PMID 25926665
- [Background] Viner RM, Christie D, Taylor V, Hey S. Motivational/solution-focused intervention improves HbA1c in adolescents with Type 1 diabetes: a pilot study. Diabet Med. 2003 Sep;20(9):739-42. doi: 10.1046/j.1464-5491.2003.00995.x. PMID 12925054
- [Background] Rosenberg AR, Yi-Frazier JP, Eaton L, Wharton C, Cochrane K, Pihoker C, Baker KS, McCauley E. Promoting Resilience in Stress Management: A Pilot Study of a Novel Resilience-Promoting Intervention for Adolescents and Young Adults With Serious Illness. J Pediatr Psychol. 2015 Oct;40(9):992-9. doi: 10.1093/jpepsy/jsv004. Epub 2015 Feb 11. PMID 25678533
- [Background] Steinhardt MA, Mamerow MM, Brown SA, Jolly CA. A resilience intervention in African American adults with type 2 diabetes: a pilot study of efficacy. Diabetes Educ. 2009 Mar-Apr;35(2):274-84. doi: 10.1177/0145721708329698. Epub 2009 Feb 9. PMID 19204102
- [Background] Maslow G, Adams C, Willis M, Neukirch J, Herts K, Froehlich W, Calleson D, Rickerby M. An evaluation of a positive youth development program for adolescents with chronic illness. J Adolesc Health. 2013 Feb;52(2):179-85. doi: 10.1016/j.jadohealth.2012.06.020. Epub 2012 Aug 17. PMID 23332482
- [Background] Schoenfeld D. Statistical considerations for pilot studies. Int J Radiat Oncol Biol Phys. 1980 Mar;6(3):371-4. doi: 10.1016/0360-3016(80)90153-4. No abstract available. PMID 7390914
- [Background] Buchanan, C. M., & Holmbeck, G. N. (1998). Measuring beliefs about adolescent personality and behavior. J. Youth Adolescence 27(5): 607-627
- [Background] Olson, D. H. Family inventories: Inventories used in a national survey of families across the life cycle. St Paul, MN: Family Social Science, University of Minnesota. 1985
- [Background] Diener, E. et al. (2010). New Well-being Measures: Short Scales to Assess Flourishing and Positive and Negative Feelings. Social Indicators Research, 97(2), 143-156.
- [Background] Walsh JC, Mandalia S, Gazzard BG. Responses to a 1 month self-report on adherence to antiretroviral therapy are consistent with electronic data and virological treatment outcome. AIDS. 2002 Jan 25;16(2):269-77. doi: 10.1097/00002030-200201250-00017. PMID 11807312
- [Background] Hair, EC et al. (2005). The Parent-Adolescent Relationship Scale. Adolescent & Family Health, 4(1), 12-25.
- [Derived] Miller VA, Silva K, Friedrich E, Robles R, Ford CA. Efficacy of a Primary Care-Based Intervention to Promote Parent-Teen Communication and Well-Being: A Randomized Controlled Trial. J Pediatr. 2020 Jul;222:200-206.e2. doi: 10.1016/j.jpeds.2020.03.050. Epub 2020 May 19. PMID 32444221